CLINICAL TRIAL: NCT02846766
Title: A Multicenter, Histology-Independent Study of the Fibroblast Growth Factor Receptor (FGFR) Inhibitor Lenvatinib (E7080) in Patients With Advanced Cancer and Aberrations in FGF/FGFR Signaling
Brief Title: Study of Lenvatinib in Patients With Advanced Cancer and Aberrations in FGF/FGFR Signaling
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to execute a contract agreement with the drug manufacturer.
Sponsor: Teresa Helsten, MD (Other)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Teresa Helsten, MD, Associate Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150659
Record Dates: First submitted 2016-05-12; First posted 2016-07-27 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Cancer
Keywords: advanced cancer; FGF; FGFR; Fibroblast Growth Factor Receptor
MeSH Terms: conditions — Neoplasms; Acrocephalosyndactylia | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenvatinib (Experimental): The starting dose of lenvatinib will be 24 mg orally per day. The duration of one cycle is defined as 28 days (4 weeks). Subjects will be treated for 2 cycles (8 weeks) and then restaged. Subjects will continue study drug until progression or unacceptable toxicity occurs.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib is administered orally at a starting dose of 24 mg per day. Lenvatinib is administered in cycles of 28 days.
  Other Names: E7080; LENVIMA

SUMMARY:
This is a two center, open label, non-randomized Phase II study of lenvatinib in adult subjects with recurrent or refractory advanced cancers with aberration(s) in FGF/FGFR signaling. Treatment will consist of daily oral administration of Lenvatinib in 28-day cycles.

DETAILED DESCRIPTION:
This exploratory, histology-independent study will enroll up to 39 subjects regardless of FGF/FGFR aberration or cancer type in order to test the hypothesis that subjects with advanced cancers harboring changes in FGF/FGFR-related genes will respond to the multikinase inhibitor lenvatinib at a higher rate than unselected cancer patients, regardless of the tumor histological subtype.

Lenvatinib is a multikinase inhibitor that inhibits FGFR1-4 as well as VEGFR1-3, RET, KIT and PDGFR-beta. It inhibits FGFR1 with an IC50 of 46 nmol/L, which is highly potent at a clinically relevant concentration.

Fibroblast growth factor (FGF) and FGF receptor (FGFR) pathway aberrations are common in malignancy, making this pathway a potentially appealing target for anti-cancer therapy. Clinical trial data suggest that targeting FGFR is indeed effective in cancer. However, the majority of such data come from trials in patient populations unselected for FGF/FGFR pathway abnormalities. The true response rates or clinical benefits for those whose cancers harbor FGF/FGFR abnormalities may be higher than observed in unselected patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Pathologically confirmed advanced or metastatic malignancy characterized by one or more of the following: Subject is intolerant of standard therapy. Malignancy is refractory to standard therapy. Malignancy relapsed after standard therapy. Malignancy for which there is no standard therapy that improves survival by at least 3 months.
* Evaluable tumor(s) with documented alteration(s) in FGF/FGFR-related gene(s). The FGF/FGFR aberration(s) can be identified at any point in the subject's cancer course. FGF/FGFR testing must have been performed in a CLIA-certified laboratory. Amplification(s) and/or mutation frequenc(ies) will be defined according to the standard of the test used. One example, Foundation OneTM, defines amplifications as ≥ 6 copies and base substitution mutations as present if there is ≥ 5% mutant allele frequency.
* Subjects must meet the following laboratory requirements at screening (may be repeated): Adequate bone marrow function: absolute neutrophil count ≥ 1,500/mL; hemoglobin ≥ 8.5 g/dL, platelets ≥ 75,000/mL. Adequate liver function: transaminases (AST/ALT) and alkaline phosphatase ≤ 3 (≤ 5 X Upper Limit of Normal (ULN) in the setting of liver metastasis) x ULN; bilirubin ≤ 1.5 x ULN. Adequate renal function: creatinine clearance ≥ 40 mL/min (Cockcroft Gault). Adequate blood coagulation: international normalized ratio (INR) ≤ 2.3. Serum amylase and lipase ≤ 1.5 x ULN.
* Adequately controlled blood pressure (BP): BP ≤ 150/90 mm Hg at screening (may be repeated and may be controlled with anti-hypertensive medication).
* Adequate performance status (PS): Eastern Cooperative Oncology Group (ECOG) PS 0-2
* Women of childbearing potential must have a negative baseline blood pregnancy test. Women and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study and for at least 30 days after discontinuation of study drug (the half life of lenvatinib is about 28 hours in patients with cancer).
* Subjects must be off other anti-tumor agents for at least 5 half lives of the agent or 4 weeks from the last day of treatment, whichever is shorter. Endocrine therapies (for example for breast or prostate cancer) and anti-Her2 therapies (for example, trastuzumab or lapatinib) are allowed to continue while on this study.
* Subjects may not be receiving any other experimental agents or agents that are not FDA approved.
* Ability to understand and willingness to sign a written consent document.

Exclusion Criteria:

* Pregnant or lactating women.
* Subjects with known hypersensitivity to any of the components or metabolites of the drug product.
* Subjects with FGFR mutations known to be inactivating. Mutations of unknown significance (based on most currently available information) will be allowed.
* Subjects who have not recovered from toxicities as a result of prior anticancer therapy, except alopecia and infertility. Recovery is defined as < Grade 2 severity per Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0).
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening.
* Inability to swallow pills or determination by the investigator that absorption of oral medication would be impaired.
* Major surgery (not including placement of central lines) within 3 weeks prior to randomization or planned surgery during the course of this study.
* Any medical condition which, in the opinion of the investigator, would preclude study participation.
* Subjects who are considered members of a vulnerable population (for example, prisoners).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rates | 2 months

SECONDARY OUTCOMES:
Clinical Benefit Rate (Complete Response, Partial Response, or Stable Disease greater than 6 months) | 6 months
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4.0 | 2 years
  Adverse events will be evaluated to determine:
  * duration (start and end dates)
  * severity (grade)
  * seriousness
  * relationship to study agent
  * action taken (i.e., none, study agent modification, medical intervention)
  * outcome (i.e., resolved without sequelae, resolved with sequelae, ongoing)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Helsten, MD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No